CLINICAL TRIAL: NCT02721888
Title: Effect of Liraglutide on Fatty Liver Content Evaluated by Proton-spectroscopy (1H-spectroscopy) and Lipoprotein Kinetic, in Patients With Type 2 Diabetes
Brief Title: Effect of Liraglutide on Fatty Liver Content and Lipoprotein Metabolism
Acronym: LIRA-NAFLD/LIP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VERGES NOVO 2012
Record Dates: First submitted 2016-02-29; First posted 2016-03-29 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Magnetic Resonance Spectroscopy; Blood Specimen Collection

ARMS (1):
- Main study (Experimental)
  Interventions: Drug: Liraglutide; Drug: MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy); Biological: Blood sample; Other: Kinetic substudy (10 patients)

INTERVENTIONS:
Drug: Liraglutide
Drug: MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy)
Biological: Blood sample
Other: Kinetic substudy (10 patients)

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is commonly associated with obesity, metabolic syndrome and type 2 diabetes. NAFLD, in patients with type 2 diabetes, has been shown to be associated with lipid abnormalities (such as hypertriglyceridemia and decreased HDL-cholesterol) and increased cardiovascular risk. Such lipid abnormalities (hypertriglyceridemia and decreased HDL-cholesterol) are very frequent in patients with type 2 diabetes. Moreover, NAFLD is a risk for further development of cirrhosis (estimated between 3 and 5%).

Animal studies have shown that liraglutide is able to decrease liver fat content, but the effect of liraglutide on liver fat content in patients with diabetes remains unknown.

In addition, human studies with liraglutide have shown significant modification of plasma lipids, such as reduction of plasma triglycerides and LDL-cholesterol. However, the mechanisms responsible for these liraglutide induced lipid modifications are not yet known.

Because increased in liver fat content and hypertriglyceridemia are associated in patients with type 2 diabetes, it seems interesting to study the effect of liraglutide on both liver fat content and lipid metabolism using gold-standard methods (proton-spectroscopy for liver fat content assessment and kinetic study with stable isotope to study lipoprotein metabolism).

This is a monocentric study. Fatty liver content will be performed by proton-spectroscopy in patients with type 2 diabetes (n=120) before and after a 6 month period of liraglutide therapy (1.2 mg/day).

Moreover, an in vivo kinetic study will be performed with stable isotopes (13C leucine) in 10 patients among the 120 patients with type 2 diabetes (n=10) before and after a 6-month period of liraglutide (1.2 mg/day) therapy. Each kinetic study will be performed during a 2-day hospitalization

For the main study, 3 visits will be performed:

* a first visit at T0, before starting the treatment with liraglutide, including clinical and biological measurements and liver fat content assessment by proton-spectroscopy
* a visit at 3 months including clinical and biological measurements
* and a visit at 6 months including clinical and biological measurements and liver fat content assessment by proton-spectroscopy

For the kinetic substudy, performed in 10 patients, a kinetic study with stable isotope will been performs during a 48h-hospitalization before starting the treatment with liraglutide and after 6 month-treatment with liraglutide

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Patients treated by metformin and/or sulfonylureas (or glinides) and/or acarbose and/or insulin,
* HbA1C >= 7 %,
* Patients who gave their written consent.

For the kinetic substudy:

* Patients who have the typical features of diabetic dyslipidemia (triglycerides >= 1.50 g/l and/or HDL<0.50 g/l [women], 0.40 g/l [men])

Exclusion Criteria:

* Treatment with thiazolidinediones or other Glucagon-like peptide-1(GLP1) agonist.
* No treatment with a Dipeptidyl peptidase-4 (DPP4) inhibitor during the 3 previous months,
* Renal or hepatic failure,
* Contra-indication for proton-spectroscopy (pacemaker, implantable prosthesis,..),
* Pregnancy.

For the kinetic substudy:

* Patients on hypolipidemic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Effect of liraglutide on fatty liver content evaluated by proton-spectroscopy (1H-spectroscopy and lipoprotein kinetics, in patients with type 2 diabetes | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Very Low Density Lipoprotein 1 (VLDL1) apolipoprotein B (apoB) production rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Very Low Density Lipoprotein 2 (VLDL2) apolipoprotein B (apoB) production rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Intermediate Density Lipoprotein (IDL) apolipoprotein B (apoB) production rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Low Density Lipoprotein (LDL) apolipoprotein B (apoB) production rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on High Density Lipoprotein (HDL) apolipoprotein A1 (apoA1) production rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Very Low Density Lipoprotein 1 (VLDL1) apolipoprotein B (apoB) fractional catabolic rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Very Low Density Lipoprotein 2 (VLDL2) apolipoprotein B (apoB) fractional catabolic rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Intermediate Density Lipoprotein (IDL) apolipoprotein B (apoB) fractional catabolic rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on Low Density Lipoprotein (LDL) apolipoprotein B (apoB) fractional catabolic rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
Effects of liraglutide on High Density Lipoprotein (HDL) apolipoprotein A1 (apoA1) fractional catabolic rate | Before and after 6 month-treatment with liraglutide (1.2 mg/day)

SECONDARY OUTCOMES:
Modification of body weight | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
  Modification of weight, induced by liraglutide 1.2 mg/d therapy.
Modification of subcutaneous fat by Magnetic Resonance Imaging (MRI) | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
  Modification of subcutaneous fat by MRI induced by liraglutide 1.2mg/d therapy
Modification of visceral fat by Magnetic Resonance Imaging (MRI) | Before and after 6 month-treatment with liraglutide (1.2 mg/day)
  Modification of visceral fat by MRI induced by liraglutide 1.2mg/d therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Result] Verges B, Duvillard L, Pais de Barros JP, Bouillet B, Baillot-Rudoni S, Rouland A, Sberna AL, Petit JM, Degrace P, Demizieux L. Liraglutide Reduces Postprandial Hyperlipidemia by Increasing ApoB48 (Apolipoprotein B48) Catabolism and by Reducing ApoB48 Production in Patients With Type 2 Diabetes Mellitus. Arterioscler Thromb Vasc Biol. 2018 Sep;38(9):2198-2206. doi: 10.1161/ATVBAHA.118.310990. PMID 30026275
- [Derived] Denimal D, Bergas V, Pais-de-Barros JP, Simoneau I, Demizieux L, Passilly-Degrace P, Bouillet B, Petit JM, Rouland A, Bataille A, Duvillard L, Verges B. Liraglutide reduces plasma dihydroceramide levels in patients with type 2 diabetes. Cardiovasc Diabetol. 2023 May 4;22(1):104. doi: 10.1186/s12933-023-01845-0. PMID 37143040
- [Derived] Verges B, Duvillard L, Pais de Barros JP, Bouillet B, Baillot-Rudoni S, Rouland A, Petit JM, Degrace P, Demizieux L. Liraglutide Increases the Catabolism of Apolipoprotein B100-Containing Lipoproteins in Patients With Type 2 Diabetes and Reduces Proprotein Convertase Subtilisin/Kexin Type 9 Expression. Diabetes Care. 2021 Apr;44(4):1027-1037. doi: 10.2337/dc20-1843. Epub 2021 Feb 2. PMID 33531418